CLINICAL TRIAL: NCT04055844
Title: A Multi-Center Phase 2 Study of Combined Modality Treatment With Ruxolitinib, Decitabine, and Donor Lymphocyte Infusion for Post-Transplant Relapse of AML or MDS
Brief Title: Multi-Ctr PII Cmb.Modality Tx Ruxolitinib, Decitabine, and DLI for Post HSCT in AML/MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018LS066; MT2018-07 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Myeloid and Monocytic Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Myelodysplastic Syndromes | interventions — Decitabine; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine + Ruxolitinib + DLI (Experimental): Eligible subjects will receive up to 4 cycles of combined modality treatment. The number of cycles depends on response, toxicity, and the remaining cell dose.
  Interventions: Drug: Decitabine; Drug: Ruxolitinib; Drug: Donor Lymphocyte Infusion (DLI)

INTERVENTIONS:
Drug: Decitabine — 10 days of decitabine 20 mg/m2 IV daily; or, alternatively, per institution, physician, or patient preference on a 5-2-5 schedule with no weekend infusion. If a CR is achieved after 2 cycles using the 10-day schedule, subsequent cycles will change to a 5-day schedule.
Drug: Ruxolitinib — Starting with day 1 of cycle 1 and continuing for up to 6 months after the end of the last cycle, patients will receive ruxolitinib 5 mg twice daily orally. Dose may be increased to 10 mg twice daily in cycles 2 through 4 if platelets improve to >100 x 10^9/L.
Drug: Donor Lymphocyte Infusion (DLI) — DLI from the original donor will be infused within 10 days after the last dose of decitabine in each cycle.

SUMMARY:
This is a multi-center, single-arm, open-label, phase II trial for the frontline treatment of relapsed AML or MDS following allo-HCT. Eligible subjects will receive up to 4 cycles of combined modality treatment. The number of cycles depends on response, toxicity, and the remaining cell dose.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥12 years
* Have undergone first allo-HCT from a 6/6 matched sibling donor, 8/8 matched unrelated donor, or an HLA haploidentical donor.
* History of AML or MDS for which allo-HCT was performed. Overlap MPN/MDS is included.
* Untreated relapse of the underlying malignancy as defined by >5% of malignant blasts (by morphology and/or flow cytometry) in the bone marrow, or myeloid sarcoma.
* Additional cells sufficient for the first DLI available from the same donor, or the donor must be willing to donate. Both G-CSF mobilized and unmobilized products are allowed and the choice is at the discretion of the treating physician.
* Partial (or better) engraftment from the bone marrow showing relapse, defined as >50% donor chimerism on non-split RFLP. Patients with chimerism of 25-50% may be enrolled with approval of the site PI and Sponsor/Investigator
* Karnofsky performance status ≥ 50%
* Adequate organ function within 14 days of study registration defined as:

  * Total bilirubin < 1.5 x upper limit of institutional normal, unless a diagnosis of Gilbert's disease
  * AST/ALT < 2.5 x upper limit of institutional normal
  * Creatinine clearance ≥40 mL/minute as calculated by the Cockcroft-Gault formula. Cockcroft-Gault CrCl = (140-age) * (Wt in kg) * (0.85 if female) / (72 * Cr).
* Peripheral white blood cell count <50 x 10^9/L. The use of hydroxyurea for cytoreduction is allowed and may continue until cycle 2 day 1
* Subjects and spouse/partner who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting at Screening and continuing through the entire study (for at least 3 months after the last dose of ruxolitinib if study treatment is stopped early or subject withdraws consent). Highly effective contraception is defined as:

  * Established use of oral, injected or implanted hormonal methods of contraception.
  * Placement of an intrauterine device or intrauterine system.
  * Double barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository (double barrier method will count as 2 forms of contraception).
* Male subjects must not donate sperm during the Screening and Treatment Periods, and for at least 3 months after the last dose of ruxolitinib.
* Subjects are willing and able to give written informed consent and to comply with all study visits and procedures. Parents or legal guardians will consent for minors and minors will be asked to assent.

Patient Exclusion Criteria:

* Active uncontrolled infection at the time of consent. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without signs or symptoms of infection will not be interpreted as an active uncontrolled infection. Subjects with a controlled infection receiving definitive therapy for 72 hours prior to enrollment are eligible.
* History of infection with human immunodeficiency virus (HIV), unresolved hepatitis B, or hepatitis C.
* Untreated CNS leukemia
* Untreated or active GVHD (acute or chronic)
* History of grade III-IV acute GVHD at any point in time
* Any form of iatrogenic immunosuppression except <0.5 mg/kg/day of prednisone or equivalent at the time of consent.
* Unresolved veno-occlusive disease of the liver, defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction (renal, ascites).
* Subjects who are pregnant, breast feeding or sexually active and unwilling to use effective birth control for the duration of the study, as agents in this study are in pregnancy category C: Animal reproduction studies have shown an adverse effect on the fetus and there are no adequate and well-controlled studies in humans, and category D: there is positive evidence of human fetal risk based on adverse reaction data from investigational or marketing experience or studies in humans.
* Radiation therapy within 14 days prior to consent.
* Any prior therapy for relapse after allo-HCT.
* Prior DLI. CD34-selected boost is allowed
* Exposure to any other investigational agent, device or procedure within 14 days prior to consent
* Patients or donors with any medical or psychological condition that, in the opinion of the Investigator, might interfere with the subject's participation in the trial, pose any additional risk for the patient/donor, or confounds the assessments of the subject.
* Subjects with known allergies, hypersensitivity or intolerance to ruxolitinib or similar compounds.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota; Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine; John F Dipersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine; Eric Huselton, M.D., Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decitabine + Ruxolitinib + DLI
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 12
Not completed — Poor Performance | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Combined Modality Treatment (Ruxolitinib, Decitabine, and DLI) for Relapsed AML or MDS Post Allo-HCT: Rate of Overall Survival (OS)
Description: Rate of Overall Survival (OS)
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 36 [18 to 72]

2. Secondary Outcome: Efficacy of Combined Modality Treatment (Ruxolitinib, Decitabine, and DLI) for Relapsed AML or MDS Post Allo-HCT: Rate of Overall Survival (OS)
Description: Rate of Overall Survival (OS)
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 14 [4 to 52]

3. Secondary Outcome: Percentage of Participants With Grade II-IV Acute Graft-versus-host Disease (aGVHD II-IV)
Description: Percentage of Participants with Grade II-IV Acute Graft-versus-host Disease (aGVHD II-IV)
Time Frame: 3 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 43 [17 to 67]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Rate of Progression Free Survival (PFS)
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants with PFS
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants with PFS | 14 [4 to 52]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Rate of Progression Free Survival (PFS)
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 7 [1 to 47]

6. Secondary Outcome: Relapse
Description: Cumulative Incidence of Relapse
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 71 [37 to 89]

7. Secondary Outcome: Relapse
Description: Cumulative Incidence of Relapse
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 79 [41 to 94]

8. Secondary Outcome: Complete Remission (CR)
Description: Rate of Complete Remission (CR)
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 14 [4 to 40]

9. Secondary Outcome: Complete Remission (CR)
Description: Rate of Complete Remission (CR)
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 7 [0 to 31]

10. Secondary Outcome: Non-Relapse Mortality (NRM)
Description: Cumulative Incidence of Non-Relapse Mortality (NRM)
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 14 [2 to 38]

11. Secondary Outcome: Non-Relapse Mortality (NRM)
Description: Cumulative Incidence of Non-Relapse Mortality (NRM)
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 14 [2 to 38]

12. Secondary Outcome: Best Response
Description: Best response until next line of treatment, death, or last follow up, whichever occurs sooner
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Decitabine + Ruxolitinib + DLI
Number analyzed (Participants) | 14
Percentage of participants | 14 [2 to 38]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Decitabine + Ruxolitinib + DLI
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Ruxolitinib + DLI (N=14)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (11)
Lung infection (Blood and lymphatic system disorders) | 1 (1)
Upper gastrointestinal (Blood and lymphatic system disorders) | 1 (2)
Alanine aminotransferase (Blood and lymphatic system disorders) | 1 (2)
Blood and lymphatic system (Cardiac disorders) | 1 (1)
Upper gastrointestinal (Cardiac disorders) | 1 (1)
Alanine aminotransferase (Cardiac disorders) | 1 (2)
Febrile neutropenia (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system (Gastrointestinal disorders) | 1 (2)
Neoplasms benign, malignant and (Gastrointestinal disorders) | 1 (1)
Sepsis (General disorders) | 1 (2)
Infections and infestations - Other, (General disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2)
Infections and infestations - Other, (Infections and infestations) | 2 (7)
Tooth infection (Infections and infestations) | 1 (1)
Intracranial hemorrhage (Infections and infestations) | 1 (1)
INR increased (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Gastrointestinal disorders - Other, (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Injury, poisoning and procedural (Infections and infestations) | 1 (1)
Alanine aminotransferase (Infections and infestations) | 1 (3)
Neoplasms benign, malignant and (Infections and infestations) | 1 (1)
Encephalopathy (Investigations) | 1 (2)
Fatigue (Investigations) | 1 (1)
General disorders and administration (Investigations) | 1 (2)
Pericardial effusion (Investigations) | 1 (3)
Syncope (Investigations) | 1 (2)
Hypertension (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Febrile neutropenia (Nervous system disorders) | 1 (2)
Sepsis (Nervous system disorders) | 1 (3)
Infections and infestations - Other, (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine + Ruxolitinib + DLI (N=14)
Bacteremia (Infections and infestations) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Hepatic infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Neutrophil count decreased (Investigations) | 8 (10)
Alanine aminotransferase increased (Investigations) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 2 (3)
INR increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (11)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hepatobiliary disorders (Cardiac disorders) | 1 (1)
Hepatic failure (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04055844/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT04055844/ICF_001.pdf